CLINICAL TRIAL: NCT00968253
Title: Phase I/II Study of Hyper-CVAD Plus RAD001 (Everolimus) for Patients With Relapsed or Refractory Acute Lymphocytic Leukemia (ALL)
Brief Title: RAD001 Study in Treatment of Relapsed or Refractory Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0100; NCI-2011-01814 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Leukemia; Acute Lymphocytic Leukemia
Keywords: Acute Lymphocytic Leukemia; ALL; Hyper-CVAD; Everolimus; 6-mercaptopurine; Citrovorum; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; G-CSF; Methotrexate; MESNA; Pegfilgrastim; Prednisone; RAD001; Solumedrol; Vincristine Sulfate
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Everolimus; Cyclophosphamide; Vincristine; Doxorubicin; Dexamethasone; Calcium Dobesilate; Mesna; Methotrexate; Cytarabine; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I: RAD001 + Combination Chemo (Experimental): Optimal dose finding of Everolimus (RAD001) beginning dose 5 mg + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Cycles 1, 3, 5, & 7 and Methotrexate & Cytarabine (Ara-C) during Cycles 2, 4, 6, & 8.
  First chemotherapy combination Hyper-CVAD = Cyclophosphamide, Vincristine, Adriamycin (doxorubicin), and Dexamethasone; Second chemotherapy combination Methotrexate and Ara-C.
  Interventions: Drug: Everolimus (RAD001); Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Mesna; Drug: Methotrexate; Drug: Ara-C (Cytarabine); Drug: Methylprednisone; Drug: G-CSF
- Phase II: MTD RAD001 + Combination Chemo (Experimental): MTD dose of Everolimus + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Cycles 1, 3, 5, & 7 and Methotrexate & Ara-C during Cycles 2, 4, 6, & 8.
  Interventions: Drug: Everolimus (RAD001); Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Dexamethasone; Drug: Mesna; Drug: Methotrexate; Drug: Ara-C (Cytarabine); Drug: Methylprednisone; Drug: G-CSF

INTERVENTIONS:
Drug: Everolimus (RAD001) — Beginning dose of 5 mg tablets every other day by mouth followed by a big glass of water. First dose will occur 1 day before receiving chemotherapy.
  Other Names: Afinitor
Drug: Cyclophosphamide — 300 mg/m^2 intravenous (IV) over 3 hours every 12 hours x 6 doses on Days 1, 2, 3 (total dose 1800 mg/m2).
  Other Names: Cytoxan; Neosar
Drug: Vincristine — 2 mg IV on Day 4 and Day 11 ± 2 days.
Drug: Doxorubicin — 50 mg/m^2 IV over 24 hours via central venous catheter on day 4, after last dose of Cyclophosphamide given.
  Other Names: Adriamycin; Rubex
Drug: Dexamethasone — 40 mg IV or orally daily days 1-4 ± 2 days and days 11-14 ± 2 days.
  Other Names: Decadron
Drug: Mesna — 600 mg/m^2 IV continuous infusion daily for 24 hours days 1-3.
  Other Names: Mesnex
Drug: Methotrexate — 200 mg/m^2 IV over 2 hours followed by 800 mg/m^2 IV over 22 hours day 1.
Drug: Ara-C (Cytarabine) — 3 gm/m^2 IV over 2 hours every 12 hours for 4 doses on days 2, 3.
  Other Names: Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Methylprednisone — 50 mg IV over 2 hours approximately every 12 hours for 6 doses days 1-3.
  Other Names: Medrol; Depo-Medrol; Solu-Medrol
Drug: G-CSF — 10 mcg/kg/day (rounded) within 72 ± 48 hours after completion of chemotherapy until neutrophil recovery 1 x 109/L or higher. Pegfilgrastim (given at 6 mg subcutaneous for one dose approximately 24 hours after completion of the chemotherapy) may be substituted for G-CSF.
  Other Names: Filgrastim; Neupogen; Granulocyte Colony Stimulating Factor

SUMMARY:
The goal of Phase I of this clinical research study is to find the highest tolerable dose of RAD001 (everolimus) when given in combination with the standard chemotherapy regimens to patients with ALL.

The goal of Phase II of this study is to learn if the drug combinations can help to control ALL. The safety of these drug combinations will be also studied in both phases.

DETAILED DESCRIPTION:
The Study Drugs:

Everolimus is designed to stop cancer cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, which may cause the tumor cells to die.

You will receive everolimus with 2 different chemotherapy combinations during alternating cycles. This means that you will receive 1 combination on Cycles 1, 3, 5, and 7 and the other combination during Cycles 2, 4, 6, and 8.

The first chemotherapy regimen is called hyper-CVAD. Hyper-CVAD includes cyclophosphamide, vincristine, Adriamycin (doxorubicin), and dexamethasone. This combination is designed to kill leukemia cells.

The other chemotherapy regimen includes the drugs methotrexate and ara-C (cytarabine). This combination is also designed to kill leukemia cells.

Study Groups and Everolimus Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 3 groups of 3-6 participants will be enrolled in the Phase I portion of the study, and up to 30 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of everolimus you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of everolimus. Each new group will receive a higher dose of everolimus than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of everolimus is found.

If you are enrolled in Phase II, you will receive everolimus at the highest dose that was tolerated in the Phase I portion.

In this study, everolimus is the only study drug where different dose levels are being tested and compared. All other drugs will be given at the same dose level.

Central Venous Catheter (CVC):

If you do not already have a CVC, you will have a CVC placed. A CVC is a plastic tube usually placed under the collarbone. You will sign a separate consent for this procedure. Some of the study drugs will be given through the CVC.

Everolimus Administration:

During all cycles, you will take everolimus once a day followed by a big glass of water. The tablets must not be chewed, broken or crushed. You may either take everolimus on an empty stomach or after a low fat meal. Taking everolimus after large, fatty meals is not advised because it will lower the amount of everolimus your body absorbs. Some examples of a low fat meal include: cereal with fat free milk, muffin/bagel with fat free spread, fruit salad, and so on. Always follow the instructions for use of everolimus given to you by your study doctor. Your first dose of everolimus will occur 1 day before you begin receiving chemotherapy.

Do not miss any tablets/capsules. You should take everolimus about the same time each day preferably in the morning.

If your study doctor thinks it is needed or if you experience severe side effects, everolimus may be stopped and then started again with a lower dose or may be stopped completely.

Chemotherapy Administration:

Each cycle will last about 21 days. The timing of each new cycle will depend on when your blood counts recover.

Cycles 1, 3, 5, and 7:

During Cycles 1, 3, 5, and 7, you will receive hyper-CVAD. The drugs will be given at the following times:

* On Days 1-3, you will receive cyclophosphamide by vein over 2-3 hours every 12 hours.
* On Days 1-4 and 11-14, you will receive dexamethasone by mouth or by vein. If by vein, the infusion will take a few seconds.
* On Day 4, you will receive doxorubicin over 24 hours through a CVC.
* On Days 4 and 11, you will receive vincristine by vein over 2-3 hours.

Cycles 2, 4, 6, and 8:

During Cycles 2, 4, 6, and 8, you will receive the methotrexate and cytarabine by vein as follows:

* On Day 1, you will receive methotrexate by vein over 24 hours.
* On Day 1, you may receive leucovorin (citrovorum) by vein (over 15 minutes) for 2-3 days. Leucovorin is given to help prevent methotrexate side effects.
* On Days 2-3, you will receive cytarabine by vein over 2 hours every 12 hours.
* On Days 1-3, you will receive methylprednisone over 2 hours every 12 hours for 6 doses.

Cycles 1-8:

You will also receive either Neupogen (filgrastim) or pegfilgrastim to help your bone marrow recover from chemotherapy. Filgrastim or pegfilgrastim will be injected under the skin within 72 hours after each cycle of chemotherapy. If you receive filgrastim, it will be given daily until your counts recover. If you receive pegfilgrastim, it will be given 1 time.

You will also receive small doses of methotrexate and Ara-C, one after the other, by a spinal tap to help prevent the disease from coming back in the fluid surrounding your brain during each cycle. During a spinal tap, a doctor or technician inserts a needle through the skin and the soft tissues of the lower back to reach a pocket of fluid that is part of the fluid space that surrounds the brain and the spinal cord. Once the fluid space is reached, chemotherapy drugs can be administered. The procedure is done under local anesthesia. An Ommaya reservoir (which holds the drugs being given) may also be implanted surgically if you have difficulty with the spinal treatments. An Ommaya reservoir is a tube inserted under the skin of the scalp that enters into the spinal fluid cavity of the brain. You will be asked to sign a separate consent form for this procedure. The number of doses you receive will depend on how many doses the study doctor thinks are needed. If you start with leukemia in the brain, it will be given 2 times a week until there is no leukemia present and then 1 time a week for 4 weeks. Sometimes, a sample of the spinal fluid collected from the spinal taps may be tested to look for leukemia cells.

Maintenance Chemotherapy:

After you have completed 8 cycles, you will begin monthly (about every 28 days, depending on your blood cell count recovery) maintenance chemotherapy for about the next 24 months. You will take the following drugs:

* You will take 6-mercaptopurine by mouth with water every day.
* You will receive methotrexate by vein (over 2 hours) or mouth every week.
* You will receive vincristine by vein over 30 minutes every 28 days.
* You will take prednisone by mouth for 5 days every month.

Study Visits:

During Cycle 1, blood (about 1 tablespoon) will be drawn for routine tests 1-3 times every week. During Cycles 2-8, blood (about 1 tablespoon) will be drawn for routine tests every 1-4 weeks.

During Cycles 1 and 2, you will have physical exam every week. After Cycle 2, you will have a physical exam every 3-4 weeks.

At Weeks 2 and 3 of Cycle 1, you will have a bone marrow aspirate to check for response. Depending on the results of the sample, this will be repeated every 1-2 weeks.

At Week 4-6 of Cycle 1, you will have a chest x-ray.

After Cycle 2 is over, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 8 teaspoons) and urine will be collected for routine tests.
* You will have a bone marrow aspirate.
* You will have a chest X-ray or computed tomography (CT) scan if needed.

If you had a positive hepatitis B test at screening, every month, blood (about 1 tablespoon) will be drawn to test the level of hepatitis B virus in your blood.

If your have risk factors and/or a positive Hepatitis C test results at screening, every month, blood (about 1 tablespoon) will be drawn to test the level of Hepatitis C virus in your blood.

Length of Study:

You may receive up to 32 cycles of study drugs. You will be taken off study early if the disease gets worse, your doctor decides it is in your best interest to stop, or you have intolerable side effects.

End-of-Study Visit:

After your last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 8 teaspoons) will be drawn for routine tests.
* You will have a bone marrow aspirate.
* If your doctor thinks it is needed, you will have a chest x-ray or CT scan.

Follow-up Visits:

You will have follow-up visits every 3 to 6 months. At these visits, the following tests and procedures will be performed:

* You will have a physical exam.
* You will have a bone marrow aspirate.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a chest x-ray.

This is an investigational study. All the chemotherapy drugs used on this study are FDA approved and commercially available for treating ALL. Everolimus is FDA approved and commercially available for the treatment of certain types of breast cancer. At this time, the combination is only being used in research.

Up to 42 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory or relapsed acute lymphocytic leukemia (ALL) or lymphoblastic lymphoma (LL). Patients expressing Philadelphia chromosome (Ph+) are eligible if they have failed a prior tyrosine kinase-containing therapy.
2. Age >/= 10 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 3.
4. Adequate liver function with serum bilirubin </= 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.5 x ULN, unless proven to be related to disease infiltration.
5. Adequate renal function with serum creatinine </= 1.5 x ULN, unless proven to be related to disease infiltration.
6. No symptomatic pulmonary disease. Forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC) and diffusion capacity of carbon monoxide (DLCO) >/= 50% of expected, corrected for hemoglobin.
7. Fasting serum cholesterol </= 300 mg/dL (or </= 7.75 mmol/L); fasting triglycerides </= 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
8. Signed informed consent.

Exclusion Criteria:

1. Systemic chemotherapy within 7 days (with the exception of hydroxyurea and/or dexamethasone) prior to starting therapy and recovered from persistent acute toxicity (> grade 1) from that therapy, unless there is evidence of rapidly progressive disease. Concurrent therapy for central nervous system (CNS) prophylaxis or treatment for CNS relapse is permitted.
2. Prior treatment with or known hypersensitivity to an mammilian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus, everolimus).
3. Major surgery within 4 weeks of start of study drug.
4. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix, or basal or squamous cell carcinomas of the skin.
5. Severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study: a. Symptomatic congestive heart failure of New York Heart Association Class III or IV. b. Unstable angina pectoris or myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia. c. Uncontrolled severe infections. d. Liver disease such as cirrhosis, or severe hepatic impairment (Child-Pugh class C).
6. continuation of #5: Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B virus (HBV) DNA and hepatitis C virus (HCV) RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
7. Known history of HIV seropositivity.
8. Impairment of gastrointestinal function of gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, malabsorption syndrome or small bowel resection).
9. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Childbearing potential is a sexually mature woman who: 1)has not undergone a hysterectomy or bilateral oophorectomy; 2)has not been naturally postmenopausal for at least 24 consecutive months. Adequate contraception must be used throughout the trial and for eight weeks after the last dose of study drug, by both sexes. (Women of child bearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of therapy.)
10. Male patient whose sexual partner(s) are women of child bearing potential who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment.
11. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
12. Patients who have developed pleural effusion while on dasatinib therapy.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 18, 2009 to March 21, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Phase I: RAD001 5 mg + Combination Chemo: Everolimus (RAD001) beginning oral dose 5 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Cytarabine (Ara-C) during Even Cycles. First chemo combo Hyper-CVAD = Cyclophosphamide 300 mg/m^2 intravenous (IV) every 12 hours x 6 doses on Days 1-3 (total dose 1800 mg/m2), Vincristine 2 mg IV on Day 4 & Day 11, Adriamycin (doxorubicin) 50 mg/m^2 IV over 24 hours Day 4, after last dose Cyclophosphamide, and Dexamethasone daily 40 mg IV or orally Days 1-4 & Days 11-14 with second Methotrexate 200 mg/m^2 IV over 2 hours followed by 800 mg/m^2 IV over 22 hours Day 1 & Ara-C 3 gm/m^2 IV every 12 hours for 4 doses Days 2, 3.
  Days 1-3, Mesna: 600 mg/m^2 IV continuous infusion daily and Methylprednisone: 50 mg IV every 12 hours for 6 doses. G-CSF: 10 mcg/kg/day within 72 after completion of chemo until neutrophil recovery 1 x 10^9/L or higher.
- Phase I: RAD001 10 mg + Combination Chemo: RAD001 oral dose 10 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Cytarabine (Ara-C) during Even Cycles. First chemo combo Hyper-CVAD = Cyclophosphamide 300 mg/m^2 intravenous (IV) every 12 hours x 6 doses on Days 1-3 (total dose 1800 mg/m2), Vincristine 2 mg IV on Day 4 & Day 11, Adriamycin (doxorubicin) 50 mg/m^2 IV over 24 hours Day 4, after last dose Cyclophosphamide, and Dexamethasone daily 40 mg IV or orally Days 1-4 & Days 11-14 with second Methotrexate 200 mg/m^2 IV over 2 hours followed by 800 mg/m^2 IV over 22 hours Day 1 & Ara-C 3 gm/m^2 IV every 12 hours for 4 doses Days 2, 3.
  Days 1-3, Mesna: 600 mg/m^2 IV continuous infusion daily and Methylprednisone: 50 mg IV every 12 hours for 6 doses. G-CSF: 10 mcg/kg/day within 72 after completion of chemo until neutrophil recovery 1 x 10^9/L or higher.
- Phase II: MTD RAD001 + Combination Chemo: RAD001 oral dose 5 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Cytarabine (Ara-C) during Even Cycles. First chemo combo Hyper-CVAD = Cyclophosphamide 300 mg/m^2 intravenous (IV) every 12 hours x 6 doses on Days 1-3 (total dose 1800 mg/m2), Vincristine 2 mg IV on Day 4 & Day 11, Adriamycin (doxorubicin) 50 mg/m^2 IV over 24 hours Day 4, after last dose Cyclophosphamide, and Dexamethasone daily 40 mg IV or orally Days 1-4 & Days 11-14 with second Methotrexate 200 mg/m^2 IV over 2 hours followed by 800 mg/m^2 IV over 22 hours Day 1 & Ara-C 3 gm/m^2 IV every 12 hours for 4 doses Days 2, 3.
  Days 1-3, Mesna: 600 mg/m^2 IV continuous infusion daily and Methylprednisone: 50 mg IV every 12 hours for 6 doses. G-CSF: 10 mcg/kg/day within 72 after completion of chemo until neutrophil recovery 1 x 10^9/L or higher.
Period: Overall Study
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo
Started | 3 | 9 | 12
Completed | 3 | 6 | 5
Not Completed | 0 | 3 | 7
Not completed — Death | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Disease Progression | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: RAD001 5 mg + Combination Chemo: RAD001 oral dose 5 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Ara-C during Even Cycles.
- Phase I: RAD001 10 mg + Combination Chemo: RAD001 oral dose 10 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Ara-C during Even Cycles.
- Phase II: MTD RAD001 + Combination Chemo: RAD001 MTD oral dose 5 mg every other day before chemo + two different chemotherapy combinations during alternating cycles, Hyper-CVAD on Odd Cycles and Methotrexate & Ara-C during Even Cycles.
- Total: Total of all reporting groups
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo | Total
Number analyzed (Participants) | 3 | 9 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 29 [24 to 52] | 24 [11 to 59] | 30 [14 to 64] | 25 [11 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 2 | 6 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose [MTD] Determination by Number of Participants With Dose Limiting Toxicity (DLT)
Description: The Maximum tolerated dose (MTD) was the highest dose level at which fewer than 2 of 6 patients developed a dose limiting toxicity (DLT) in the first two cycles of therapy. A 3 by 3 design was used for dose escalation in the phase I portion of the study.
  A dose-limiting toxic effect (DLT) was defined as a clinically significant adverse event or abnormal laboratory value directly attributable to everolimus and assessed as unrelated to disease progression, intercurrent illness, or concomitant medications, occurring during the first or second cycle of therapy, that met any of the following criteria: CTCAE version 3.0 grade 3 increased AST or ALT for 7 days, CTCAE grade 4 increased AST or ALT of any duration, or any other clinically significant CTCAE grade 3 or 4 toxic effect. Electrolyte abnormalities (changes in glucose, chemistries, liver enzymes, pancreatic enzymes) correctable by optimal therapy and without clinical impact were not considered DLTs.
Time Frame: Following first two dose cycles (21 days/each), up to 42 days
Population: Maximum tolerated dose was an outcome measure for the phase I portion of this study only. MTD was already established, therefore, not analyzed on the participants for the phase II portion of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo
Number analyzed (Participants) | 3 | 6 | 0
Participants | 0 | 1 |
Statistical Analysis 1: Comparison: Phase I: RAD001 5 mg + Combination Chemo vs Phase I: RAD001 10 mg + Combination Chemo; Test type: Superiority or Other; Maximum tolerated dose = 5 — Maximum tolerated dose (MTD) of Everolimus measured in mg/day in combination with HyperCVAD

2. Primary Outcome: Overall Response Rate (OR) Where OR = CR + CRp + CRi
Description: Number of participants out of total treated who experienced a complete response response according to RECIST criteria either (CR + CRp) CR Without Platelet Recovery. Response (CR + CRp) defined as Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x10^9/L, platelet count > 100 x10^9/L, and blasts < 5% in a normocellular or hypercellular marrow. Complete remission without platelet recovery (CRp): Peripheral blood and marrow parameters as for CR, but with platelet count > 20 x 10^9/L and < 100 x 10^9/L in the absence of platelet transfusions. CR with incomplete blood count recovery (CRi): Same as CR but platelets ≤ 100,000/mcl and/or neutrophils ≤ 1,000/mcl.
Time Frame: 8 courses of treatment, up to 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo
Number analyzed (Participants) | 3 | 9 | 12
percentage of participants | 33 | 33 | 33

3. Secondary Outcome: Participant Responses by Daily Dose Level Assignment (RAD001 5 mg, 10 mg and MTD 5 mg)
Description: Response defined as Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x10^9/L, platelet count > 100 x10^9/L, and blasts < 5% in a normocellular or hypercellular marrow. Complete remission without platelet recovery (CRp): Peripheral blood and marrow parameters as for CR, but with platelet count > 20 x 10^9/L and < 100 x 10^9/L in the absence of platelet transfusions. CR with incomplete blood count recovery (CRi): Same as CR but platelets ≤ 100,000/mcl and/or neutrophils ≤ 1,000/mcl. Partial remission (PR): Peripheral blood count recovery as for CR, with decrease in marrow blasts by > 50% from pretreatment values with no more than 25% leukemia/lymphoma cells in the marrow. Nonresponder, Other: All other responses will be considered failures.
Time Frame: Up to 20 cycles of study drugs (21 day cycles) or till disease progression
Measure: Number; unit: participants
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo
Number analyzed (Participants) | 3 | 9 | 12
participants
  Complete Remission | 1 | 2 | 3
  Complete Remission without platelet recovery | 0 | 0 | 1
  CR with incomplete blood count recovery | 0 | 1 | 0
  Partial Remission | 1 | 1 | 0
  Nonresponder | 1 | 5 | 8

ADVERSE EVENTS:
Time Frame: Adverse event collection for 8 courses of trial (21 day course), up to 24 weeks; SAEs reported from time consent is signed, during the course of treatment and within 30 days after the last day of active treatment.
Arm/Group | Phase I: RAD001 5 mg + Combination Chemo | Phase I: RAD001 10 mg + Combination Chemo | Phase II: MTD RAD001 + Combination Chemo
Serious Adverse Events (participants affected / at risk) | 1/3 | 7/9 | 11/12
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: RAD001 5 mg + Combination Chemo (N=3) | Phase I: RAD001 10 mg + Combination Chemo (N=9) | Phase II: MTD RAD001 + Combination Chemo (N=12)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (10)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Infection - E Coli Bacterium (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Multi-Organ Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2) | 3 (3)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal pain, Bladder Spasms
Mucositis/Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase I: RAD001 5 mg + Combination Chemo (N=3) | Phase I: RAD001 10 mg + Combination Chemo (N=9) | Phase II: MTD RAD001 + Combination Chemo (N=12)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (7) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (10) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (7) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 6 (8)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 4 (8)
Blood/Bone Marrow (Other) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) — Epistaxis
Cardiac General (Other) (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) — cardiomyopathy, tachycardia
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Constitutional Symptoms (Other) (General disorders) | 0 (0) | 1 (1) | 0 (0) — sore mouth
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 3 (3)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Dental prosthesis, soreness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Edema limbs (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 7 (9)
Fever (General disorders) | 2 (2) | 4 (6) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (5) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/Bleeding (Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2)
Infection (Other) (Infections and infestations) | 0 (0) | 4 (4) | 6 (10) — Bacteria, Acremonium fungemia
Infection (Other) (Infections and infestations) | 0 (0) | 5 (11) | 6 (9) — ESCHERICHIA COLI, STENOTROPHOMONAS, HERPES
Infectious colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3)
Metabolic/Laboratory (Other) (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (1) — Elevated amylase and lipase
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 6 (8) | 5 (8)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) — Bilateral Edema
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pain (Other) (General disorders) | 0 (0) | 1 (1) | 0 (0) — Left Flank
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 4 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0/0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (5)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6)
Hypernatremia (Metabolism and nutrition disorders) | 0/0 (0) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0/0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes